CLINICAL TRIAL: NCT01456169
Title: A Phase-3 Randomized, Double-Blind, Efficacy and Safety Study Evaluating the Fixed Dose Combinations of TAK-491 Plus Chlorthalidone (40/12.5 mg and 40/25 mg) in Subjects With Grades 2 or 3 Essential Hypertension, Who Do Not Achieve Target Blood Pressure Following Treatment With TAK-491 40 mg Monotherapy
Brief Title: A Study to Evaluate the Effectiveness and Safety of a Fixed Dose Combination of Azilsartan Medoxomil and Chlorthalidone in Patients With High Blood Pressure Who do Not Achieve Target Blood Pressure Following Treatment With Azilsartan Medoxomil Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-491CLD_307; 2011-000220-16 (EudraCT Number); U1111-1119-4743 (Registry Identifier: WHO); 11-028 (Registry Identifier: ROCTR); NL36272.072.11 (Registry Identifier: CCMO)
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: Essential Hypertension
Keywords: High Blood Pressure; Drug Therapy
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — azilsartan medoxomil; azilsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azilsartan medoxomil 40 mg (Active Comparator): Azilsartan medoxomil 40 mg and placebo to chlorthalidone combination tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Azilsartan medoxomil/placebo
- Azilsartan medoxomil + chlorthalidone 40/12.5 mg (Experimental): Azilsartan 40 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Azilsartan medoxomil - chlorthalidone
- Azilsartan medoxomil + chlorthalidone 40/25 mg (Experimental): Azilsartan medoxomil 40 mg and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Azilsartan medoxomil - chlorthalidone

INTERVENTIONS:
Drug: Azilsartan medoxomil/placebo — Azilsartan medoxomil and placebo to chlorthalidone combination tablets
  Other Names: TAK-491; EDARBI
  Arms: Azilsartan medoxomil 40 mg
Drug: Azilsartan medoxomil - chlorthalidone — Azilsartan medoxomil and chlorthalidone fixed dose combination tablets
  Other Names: TAK-491CLD; Edarbyclor
  Arms: Azilsartan medoxomil + chlorthalidone 40/12.5 mg; Azilsartan medoxomil + chlorthalidone 40/25 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the fixed dose combinations of azilsartan medoxomil plus chlorthalidone (40/12.5 and 40/25 mg), once daily, in participants with grades 2 or 3 essential hypertension who do not reach target blood pressure following treatment with 40 mg azilsartan medoxomil monotherapy after 4 weeks.

DETAILED DESCRIPTION:
Eligible participants completed a 2-week single-blind run-in period (Days -42 to -29) prior to a Single-Blind Monotherapy Treatment Period (Day -28 to Day -1) where they received azilsartan medoxomil 40 mg. After the Single-Blind Monotherapy Treatment Period, those participants who achieved target blood pressure discontinued treatment and resumed standard of care management at the discretion of their treating physician, while those participants who did not achieve target blood pressure (defined as clinic systolic blood pressure ≥140 mmHg) were randomly assigned to 1 of 3 active treatment arms: azilsartan medoxomil 40 mg plus placebo, azilsartan medoxomil plus chlorthalidone 40/12.5 mg, or azilsartan medoxomil plus chlorthalidone 40/25 mg.

ELIGIBILITY:
Inclusion Criteria:

At Screening

1. The participant has grade 2-3 essential hypertension which is not adequately controlled, as defined by mean, trough, sitting, clinic systolic blood pressure (SBP):

   * ≥160 to ≤180 mm Hg in participants who have not received any antihypertensive medication in the 14 days prior to Visit 1.
   * ≥150 to ≤170 mm Hg in participants taking 1 antihypertensive medication at Visit 1.
   * ≥140 to ≤160 mm Hg in participants taking 2 antihypertensive medications at Visit 1.
2. The participant has clinical laboratory test results (clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory or the investigator does not consider the results to be clinically relevant for precluding entry in to the study in this hypertensive population.
3. The participant is willing to discontinue current antihypertensive medications.
4. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
5. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
6. Male or female adult, at least 18 years of age.
7. A female of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of the informed consent through 30 days after the last study drug dose. NOTE: Women NOT of childbearing potential are defined as those who have been surgically sterilized (hysterectomy, bilateral oophorectomy, tubal ligation [performed more than one 1 year prior to Screening]) or who are postmenopausal (defined as at least 1 year since last regular menses).

   Post-placebo run-in:
8. The participant must have a post-placebo run-in, 24-hour mean SBP by ambulatory blood pressure monitoring (ABPM) of 140-175 mm Hg inclusive, and a clinic SBP measurement of 160 to 190 mm Hg inclusive (determined by the mean of 3 sitting, trough, measurements on Day -29) to qualify for entry in to the 4 week single-blind TAK-491 40 mg monotherapy treatment period.

   Post-4 week, single-blind TAK-491 40 mg monotherapy treatment:
9. The participant does not achieve target blood pressure (defined as clinic SBP ≥140 mm Hg as determined by the mean of 3 sitting, trough, measurements) following 4 weeks single-blind treatment with TAK-491 40 mg monotherapy at Day -1, prior to randomization to double-blind treatment.

Exclusion Criteria:

At Screening

1. The participant has clinic diastolic blood pressure (DBP) >110 mm Hg.
2. The participant's 3 SBP measurements differ by more than 15 mm Hg (confirmed by a second set of three measurements).
3. The participant has received any investigational compound within 30 days prior to Screening or is currently participating in another investigational study. NOTE: Participants participating in observational studies (per local definition) may enter Screening provided that the last intervention or invasive procedure was >30 days prior to Visit 1.
4. The participant has been randomized/enrolled in a previous TAK-491 or TAK-491CLD study. NOTE: This criterion does not apply to participants who entered screening or placebo run-in in another TAK-491 or TAK-491CLD study but were not randomized/enrolled.
5. The participant is a study site employee or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
6. The participant is currently treated with more than 2 antihypertensive medications.
7. The participant works a night (third) shift (defined as 11 PM [2300] to 7 AM [0700]).
8. The participant has an upper arm circumference <24 cm or >42 cm.
9. The participant has secondary hypertension of any etiology (e.g., renovascular disease, pheochromocytoma, Cushing's syndrome).
10. The participant has any history of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, persistent or permanent atrial fibrillation or transient ischemic attack.
11. The participant has clinically significant cardiac conduction defects (e.g., third-degree atrioventricular block, sick sinus syndrome).
12. The participant has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease or hypertrophic cardiomyopathy.
13. The participant has severe renal dysfunction or disease [based on estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m^2 at screening], prior renal transplantation or nephrotic syndrome (defined as a urinary albumin/creatinine ratio >2000 mg/g at Screening).
14. Participant has known hemodynamically significant bilateral renal artery stenosis or unilateral disease in a single kidney.
15. The participant has a history of cancer that has not been in remission for at least 5 years prior to the first dose of single-blind TAK-491 monotherapy study drug. (This criterion does not apply to those participants with basal cell or Stage 1 squamous cell carcinoma of the skin).
16. The participant has poorly-controlled type 1 or 2 diabetes mellitus (hemoglobin A1c [HbA1c] >8.5%) at Screening.
17. The participant has hypokalemia or hyperkalemia (defined as serum potassium outside of the normal reference range of the central laboratory) at Screening.
18. The participant has an alanine aminotransferase or aspartate aminotransferase level >2.5 times the upper limit of normal, active liver disease, or jaundice at Screening.
19. The participant has any other known serious disease or condition that would compromise safety, might affect life expectancy, or make it difficult to successfully manage and follow the participant according to the protocol.
20. The participant has a history of hypersensitivity or allergies to angiotensin II receptor blockers (ARB) or thiazide-type diuretics or other sulfonamide-derived compounds.
21. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse per local guidelines within the past 2 years.
22. The participant is required to take excluded medications at any point during the study.
23. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.

    Post-placebo run-in period
24. The participant has a clinic SBP >190 mm Hg and DBP >115 mm Hg.
25. The participant is noncompliant (<70% or >130%) with study medication during the placebo run-in period.
26. The participant has a 24-hour mean eligibility ABPM reading of insufficient quality.

    Post-single-blind TAK-491 40 mg treatment period
27. The participant has a clinic SBP >180 mm Hg and DBP >110 mm Hg.
28. The participant is noncompliant (<70% or >130%) with study medication during the TAK-491 40 mg single-blind treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (108):
- Bulgaria (7):
  - Haskovo
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
  - Veliko Tarnovo
- Estonia (5):
  - Paide
  - Saku
  - Tallinn
  - Tartu
  - Võru
- France (6):
  - Labarthe-sur-Lèze, Haute Garonne
  - Bourg-des-Comptes, Ille et Vilaine
  - Tours, Indre et Loire
  - Vourey, Isere
  - Saint-Étienne-de-Montluc, Pays de la Loire Region
  - Orthez, Pyrenees Atlantiques
- Germany (10):
  - Karlsruhe, Baden-Wurttemberg
  - Bad Wörishofen, Bavaria
  - Nuremberg, Bavaria
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Stuhr, Lower Saxony
  - Essen, North Rhine-Westphalia
  - Kamp-Lintfort, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
- Hungary (8):
  - Budapest
  - Debrecen
  - Gyöngyös
  - Gyula
  - Mosonmagyaróvár
  - Nyíregyháza
  - Pécs
  - Szikszó
- Italy (13):
  - Torrette Di Ancona, Ancona
  - Acquaviva delle Fonti, Bari
  - Brescia, Brescia
  - Ferrara, Ferrara
  - L’Aquila, L'Aquila
  - Milan, Milano
  - Palermo, Palermo
  - Pavia, Pavia
  - Pisa, Pisa
  - Roma, Roma
  - Sassari, Sassari
  - Legnago, Verona
  - Bologna
- Lithuania (2):
  - Alytus
  - Kaunas
- Netherlands (10):
  - Beek
  - Breda
  - Eindhoven
  - Groningen
  - Leiderdorp
  - Maastricht
  - Rotterdam
  - Velp
  - Zoetermeer
  - Zwijndrecht
- Poland (14):
  - Bydgoszcz
  - Gdansk
  - Gdynia
  - Krakow
  - Lodz
  - Lublin
  - Oświęcim
  - Parczew
  - Poznan
  - Pulway
  - Rzeszów
  - Sopot
  - Torun
  - Zgierz
- Serbia (6):
  - Belgrade
  - Kamenitz
  - Kragujevac
  - Kruševac
  - Niš
  - Zemun
- Slovakia (12):
  - Bardejov
  - Bratislava
  - Galanta
  - Komárno
  - Košice
  - Lučenec
  - Martin
  - Nitra
  - Nové Zámky
  - Prešov
  - Svidník
  - Žilina
- Spain (4):
  - Barcelona, Barcelona
  - Centelles, Barcelona
  - Madrid, Madrid
  - Málaga, Malaga
- Sweden (4):
  - Gothenburg
  - Lund
  - Malmo
  - Vällingby
- United Kingdom (7):
  - London, Greater London
  - Glasgow, Lanarkshire
  - Blackpool, Lancashire
  - Northwood, Middlesex
  - Bath, Somerset
  - Royal Leamington Spa, Warwickshire
  - Westbury, Wiltshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1754 patients were screened at 125 investigative sites in Bulgaria, Estonia, France, Germany, Hungary, Italy, Lithuania, the Netherlands, Poland, Serbia, Slovakia, Spain, Sweden, and the United Kingdom from 31 October 2011 to 24 January 2013.
Pre-assignment Details: 507 participants entered the azilsartan medoxomil 40 mg Single-Blind Monotherapy Treatment Period and 395 participants were eligible to enter the Double-Blind Treatment Period and were randomly assigned to 1 of 3 active treatment arms.
Groups:
- Azilsartan Medoxomil 40 mg: Azilsartan medoxomil 40 mg and chlorthalidone placebo combination tablets, orally, once daily for up to 8 weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Started | 133 (Indicates participants who were randomized into the double-blind treatment period) | 127 (Indicates participants who were randomized into the double-blind treatment period) | 135 (Indicates participants who were randomized into the double-blind treatment period)
Completed | 123 | 122 | 123
Not Completed | 10 | 5 | 12
Not completed — Adverse Event | 1 | 2 | 7
Not completed — Major Protocol Deviation | 3 | 2 | 3
Not completed — Voluntary Withdrawal | 3 | 0 | 2
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Other | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were randomized into the double-blind treatment period. Baseline was defined as the last observed value while on monotherapy study drug and before the first dose of double-blind study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg | Total
Number analyzed (Participants) | 133 | 127 | 135 | 395
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.18) | 59.2 (10.72) | 57.7 (10.46) | 58.2 (10.45)
Age, Customized [Number; unit: participants]
  < 45 years | 13 | 10 | 12 | 35
  45 to < 65 years | 87 | 79 | 88 | 254
  ≥ 65 years | 33 | 38 | 35 | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 54 | 44 | 144
  Male | 87 | 73 | 91 | 251
Race/Ethnicity, Customized [Number; unit: participants] — Participants could choose more than 1 category for race and those who indicated more than 1 race category were included in each category and in the Multiracial category. Thus the total number of participants may not generally add up to the total number of each group.
  participants
    American Indian or Alaska Native | 1 | 0 | 1 | 2
    Asian | 0 | 1 | 0 | 1
    Black or African American | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
    White | 132 | 126 | 134 | 392
    Multiracial | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Bulgaria | 11 | 10 | 11 | 32
  Estonia | 18 | 16 | 18 | 52
  France | 2 | 1 | 2 | 5
  Germany | 29 | 29 | 28 | 86
  Hungary | 10 | 9 | 10 | 29
  Italy | 6 | 4 | 5 | 15
  Lithuania | 5 | 4 | 6 | 15
  Netherlands | 4 | 6 | 5 | 15
  Poland | 17 | 18 | 17 | 52
  Serbia | 4 | 3 | 4 | 11
  Slovakia | 24 | 24 | 26 | 74
  Spain | 1 | 1 | 1 | 3
  Sweden | 1 | 2 | 1 | 4
  United Kingdom | 1 | 0 | 1 | 2
Weight [Mean (Standard Deviation); unit: kg] | 87.59 (15.794) | 86.71 (17.037) | 87.39 (14.876) | 87.24 (15.868)
Height [Mean (Standard Deviation); unit: cm] — Height data only available for 126 participants in the Azilsartan medoxomil + chlorthalidone 40/12.5 mg treatment group.
  cm | 171.8 (8.87) | 170.6 (9.96) | 172.1 (9.74) | 171.5 (9.53)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI data only available for 126 participants in the Azilsartan medoxomil + chlorthalidone 40/12.5 mg treatment group.
  kg/m^2 | 29.63 (5.066) | 29.78 (5.206) | 29.52 (4.572) | 29.64 (4.937)
Smoking Classification [Number; unit: participants]
  Never smoked | 77 | 83 | 77 | 237
  Current smoker | 31 | 25 | 30 | 86
  Ex-smoker | 25 | 19 | 28 | 72
Diabetes Status [Number; unit: participants]
  Yes | 20 | 27 | 20 | 67
  No | 113 | 100 | 115 | 328
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 84.8 (16.41) | 81.5 (16.25) | 82.4 (16.51) | 82.9 (16.41)
Baseline eGFR Categories (mL/min/1.73 m^2) [Number; unit: participants]
  30 to < 60 ml/min/1.73 m^2 | 11 | 10 | 11 | 32
  60 to < 90 ml/min/1.73 m^2 | 78 | 85 | 80 | 243
  ≥ 90 ml/min/1.73 m^2 | 44 | 32 | 44 | 120
Trough Clinic Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 150.7 (10.69) | 149.6 (11.54) | 149.8 (10.95) | 150.0 (11.04)
Trough Clinic SBP Category (mmHg) [Number; unit: participants]
  <140 mmHg | 16 | 17 | 17 | 50
  ≥140 - <160 mmHg | 86 | 87 | 93 | 266
  ≥160 - <180 mmHg | 31 | 23 | 25 | 79
  ≥180 mmHg | 0 | 0 | 0 | 0
Trough Clinic Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 89.8 (7.76) | 87.6 (9.31) | 88.8 (7.99) | 88.7 (8.39)
Trough Clinic DBP Categories (mmHg) [Number; unit: participants]
  <90 mmHg | 68 | 72 | 70 | 210
  ≥90 mmHg | 65 | 55 | 65 | 185

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Trough, Sitting, Clinic Systolic Blood Pressure
Description: The change between trough systolic blood pressure measured at final visit or Week 8 relative to baseline. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline (of the double-blind treatment period) and Week 8
Population: Full analysis set, consisting of all randomized participants who received at least 1 dose of double-blind study drug. A participant was included in the analyses only when there was both a baseline value and at least 1 value during the double-blind treatment period. Last observation carried forward (LOCF) was used.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 133 | 126 | 135
mm Hg
  Baseline | 150.7 (0.96) | 149.8 (0.98) | 149.8 (0.95)
  Change from Baseline to Week 8 | -6.4 (1.05) | -15.8 (1.08) | -21.1 (1.04)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg vs Azilsartan Medoxomil + Chlorthalidone 40/25 mg; The type I error was controlled using a 2-step hierarchical testing procedure. In the first step, the high dose (40/25 mg) of Azilsartan medoxomil + chlorthalidone was compared to Azilsartan medoxomil alone. If the comparison in step 1 was statistically significant at a significance level of 5%, then step 2 was performed by comparing the low dose (40/12.5 mg) and monotherapy at the 5% significance level; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with treatment as a fixed effect and baseline trough, sitting, clinic SBP as a covariate; LS mean difference = -14.7, 95% CI 2-sided [-17.6 to -11.8]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg vs Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with treatment as a fixed effect and baseline trough, sitting, clinic SBP as a covariate; LS mean difference = -9.5, 95% CI 2-sided [-12.4 to -6.5]

2. Secondary Outcome: Change From Baseline to Week 8 in Trough, Sitting, Clinic Diastolic Blood Pressure
Description: The change between trough diastolic blood pressure measured at final visit or week 8 relative to baseline Diastolic blood pressure is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 8
Population: Full analysis set; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 133 | 126 | 135
mm Hg
  Baseline | 89.8 (0.73) | 87.7 (0.75) | 88.8 (0.72)
  Change from Baseline to Week 8 | -3.2 (0.65) | -7.7 (0.67) | -10.3 (0.65)

3. Secondary Outcome: Change From Baseline to Week 8 in Trough Systolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in trough systolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 8, 22-24 hours after dosing
Population: Full analysis set. Only participants with a baseline and at least 1 post-baseline value of acceptable quality were included.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 107 | 98 | 104
mm Hg
  Baseline | 143.1 (1.55) | 140.2 (1.62) | 142.0 (1.58)
  Change from Baseline to Week 8 | -2.5 (1.31) | -14.0 (1.36) | -16.6 (1.32)

4. Secondary Outcome: Change From Baseline to Week 8 in Trough Diastolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in trough diastolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 8, 22-24 hours after dosing
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 107 | 98 | 104
mm Hg
  Baseline | 86.4 (1.11) | 83.6 (1.16) | 86.0 (1.12)
  Change from Baseline to Week 8 | -2.2 (0.88) | -8.8 (0.92) | -9.4 (0.89)

5. Secondary Outcome: Change From Baseline to Week 8 in the 24-hour Mean Systolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in 24-hour mean systolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 107 | 98 | 104
mm Hg
  Baseline | 138.0 (1.21) | 137.0 (1.26) | 138.2 (1.22)
  Change from Baseline to Week 8 | -2.3 (1.02) | -14.7 (1.07) | -18.1 (1.03)

6. Secondary Outcome: Change From Baseline to Week 8 in the 24-hour Mean Diastolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in 24-hour mean diastolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 107 | 98 | 104
mm Hg
  Baseline | 81.9 (0.89) | 80.3 (0.93) | 82.5 (0.91)
  Change from Baseline to Week 8 | -1.6 (0.66) | -8.5 (0.69) | -10.1 (0.67)

7. Secondary Outcome: Change From Baseline to Week 8 in the Mean Daytime Systolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in daytime (6 am to 10 pm) mean systolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 107 | 98 | 104
mm Hg
  Baseline | 141.5 (1.24) | 141.1 (1.30) | 141.9 (1.26)
  Change from Baseline to Week 8 | -2.4 (1.09) | -15.3 (1.14) | -18.2 (1.11)

8. Secondary Outcome: Change From Baseline to Week 8 in the Mean Daytime Diastolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in daytime (6 am to 10 pm) mean diastolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 107 | 98 | 104
mm Hg
  Baseline | 84.9 (0.96) | 83.6 (1.01) | 85.7 (0.98)
  Change from Baseline to Week 8 | -1.7 (0.72) | -8.9 (0.75) | -10.1 (0.73)

9. Secondary Outcome: Change From Baseline to Week 8 in the Mean Nighttime Systolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in nighttime (12 am to 6 am) mean systolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 107 | 98 | 104
mm Hg
  Baseline | 127.3 (1.50) | 124.2 (1.57) | 126.3 (1.52)
  Change from Baseline to Week 8 | -2.2 (1.18) | -12.7 (1.24) | -17.3 (1.20)

10. Secondary Outcome: Change From Baseline to Week 8 in the Mean Nighttime Diastolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in nighttime (12 am to 6 am) mean diastolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 8.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 107 | 98 | 104
mm Hg
  Baseline | 73.2 (0.95) | 70.6 (0.99) | 72.9 (0.97)
  Change from Baseline to Week 8 | -1.6 (0.78) | -7.2 (0.82) | -9.8 (0.79)

11. Secondary Outcome: Change From Baseline to Week 8 in the Mean Systolic Blood Pressure 0 to 12 Hours After Dosing, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in the 12-hour mean systolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 107 | 98 | 104
mm Hg
  Baseline | 141.6 (1.30) | 141.8 (1.36) | 142.3 (1.32)
  Change from Baseline to Week 8 | -2.3 (1.14) | -15.4 (1.19) | -18.2 (1.16)

12. Secondary Outcome: Change From Baseline to Week 8 in the Mean Diastolic Blood Pressure 0 to 12 Hours After Dosing, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in the 12-hour mean diastolic blood pressure measured at final visit or Week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 107 | 98 | 104
mm Hg
  Baseline | 85.2 (1.01) | 84.2 (1.05) | 86.0 (1.02)
  Week 8 | -1.6 (0.75) | -8.9 (0.78) | -10.1 (0.76)

13. Secondary Outcome: Percentage of Participants Who Achieve a Target Clinic Systolic Blood Pressure at Week 8
Description: Percentage of participants who achieve a target clinic systolic blood pressure measured at final visit or week 8, defined as less than 140 mm Hg (or less than 130 mm Hg for participants with diabetes or chronic kidney disease). Systolic blood pressure is the arithmetic mean of the 3 trough sitting Systolic blood pressure measurements.
Time Frame: Week 8
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 133 | 126 | 135
percentage of participants | 35.3 | 62.7 | 77.8

14. Secondary Outcome: Percentage of Participants Who Achieve a Target Clinic Diastolic Blood Pressure at Week 8
Description: Percentage of participants who achieve a target clinic diastolic blood pressure measured at final visit or week 8, defined as less than 90 mm Hg (or less than 80 mm Hg for participants with diabetes or chronic kidney disease). Diastolic blood pressure is based on the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Time Frame: Week 8
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 133 | 126 | 135
percentage of participants | 60.2 | 81.0 | 85.9

15. Secondary Outcome: Percentage of Participants Who Achieve Both Clinic Systolic and Diastolic Blood Pressure Targets at Week 8
Description: Percentage of participants who achieve both clinic systolic and diastolic blood pressure targets at Week 8, defined as less than 140 mm Hg (or less than 130 mm Hg for participants with diabetes or chronic kidney disease) for systolic AND less than 90 mm Hg (or less than 80 mm Hg for participants with diabetes or chronic kidney disease) for diastolic blood pressure.
Time Frame: Week 8
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Number analyzed (Participants) | 133 | 126 | 135
percentage of participants | 30.8 | 59.5 | 74.1

ADVERSE EVENTS:
Time Frame: For 4 weeks during the monotherapy treatment period and from the first dose of double-blind study drug up to 14 days (or 30 days for a Serious AE) after the last dose of study drug in the 8-week double-blind treatment period.
Description: The investigator documented any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of relation to study drug.
Groups:
- Monotherapy: Azilsartan Medoxomil 40 mg: Azilsartan medoxomil 40 mg and chlorthalidone placebo combination tablets, orally, once daily for 4 weeks during the Single-Blind Monotherapy Treatment Period. All enrolled participants, including those who were not randomized to double-blind treatment are included in this group.
- Azilsartan Medoxomil 40 mg: Azilsartan medoxomil 40 mg and chlorthalidone placebo combination tablets, orally, once daily for up to 8 weeks during the Double-Blind Treatment Period.
- Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg: Azilsartan 40 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for up to 8 weeks during the Double-Blind Treatment Period.
- Azilsartan Medoxomil + Chlorthalidone 40/25 mg: Azilsartan medoxomil 40 mg and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks during the Double-Blind Treatment Period.
Arm/Group | Monotherapy: Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg | Azilsartan Medoxomil + Chlorthalidone 40/25 mg
Serious Adverse Events (participants affected / at risk) | 3/507 | 2/133 | 0/127 | 0/135
Other Adverse Events (participants affected / at risk) | 15/507 | 15/133 | 13/127 | 26/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy: Azilsartan Medoxomil 40 mg (N=507) | Azilsartan Medoxomil 40 mg (N=133) | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg (N=127) | Azilsartan Medoxomil + Chlorthalidone 40/25 mg (N=135)
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy: Azilsartan Medoxomil 40 mg (N=507) | Azilsartan Medoxomil 40 mg (N=133) | Azilsartan Medoxomil + Chlorthalidone 40/12.5 mg (N=127) | Azilsartan Medoxomil + Chlorthalidone 40/25 mg (N=135)
Nasopharyngitis (Infections and infestations) | 6 | 4 | 2 | 4
Viral infection (Infections and infestations) | 0 | 4 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 4 | 4 | 11
Headache (Nervous system disorders) | 9 | 2 | 3 | 5
Dizziness (Nervous system disorders) | 3 | 0 | 2 | 6
Hypotension (Vascular disorders) | 0 | 1 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.